CLINICAL TRIAL: NCT06007534
Title: Caractérisation de la pharmacocinétique d'Une Dose Unique de 200 mg de Doxycycline en Prophylaxie Post-exposition (PEP) Des Infections Sexuellement Transmissibles Dans différents Compartiments Biologiques
Brief Title: Pharmacokinetic Characterization of a Single 200 mg Dose of Doxycycline in Post-exposure Prophylaxis (PEP) of Sexually Transmitted Infections in Different Biological Compartments
Acronym: DOXY-PK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP221156
Record Dates: First submitted 2023-06-30; First posted 2023-08-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Post-exposure Prophylaxis; Sexually Transmitted Diseases; Doxycycline
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult male patient (Other): Men having Sex with Men on PrEP (pre-Exposition Prophylaxy) regularly taking doxycycline for Sexually Transmitted Infection (STI) prevention or HIV-infected
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — Blood samples, urine samples and oropharyngeal swabs before taking 200mg of doxycycline and then 2h, 24h, 48h, 7 days, 14 days, 60 days and 90 days after the single dose of doxycycline Hair samples: at the time of doxycycline administration, 1 month and 3 months after the single dose of doxycycline

SUMMARY:
Post-exposure prophylaxis (PEP) using doxycycline 200 mg within 24 hours of unprotected sexual intercourse to prevent sexually transmitted infections has demonstrated a reduction in the incidence of chlamydial and syphilis infections and syphilis infection by 70% and 73% in men who have sex with men (MSM) undergoing pre-exposure prophylaxis prophylaxis (PrEP) for HIV. Other studies are underway or in development on doxycycline prophylaxis for bacterial STIs, which are particularly common in this population. Monitoring adherence to PEP is of great interest in guaranteeing the effectiveness of this strategy and to be able to assess the uptake of PEP among PrEP users. Among the many methods for assessing adherence, measuring drug concentrations is a more accurate measure of adherence than self-reporting.

The therapeutic monitoring of doxycycline and the assessment of adherence have been described using plasma and hair samples, allowing estimation of intake over the last 3-4 days and 4 months, respectively. Nevertheless, these biological matrices present several limitations for application in clinical practice: reflecting the duration of exposure should be more in line with the frequency of visits (2 months), and the collection of hair samples may be difficult due to refusal or short hair. On the other hand, interpretation of the hair assay is limited by the degradation of doxycycline in this matrix, which could lead to underestimation of drug intake. By Therefore, new biological matrices are needed for more accurate assessment of doxycycline adherence in post-exposure prevention monitoring.

The objective is to evaluate the pharmacokinetics of doxycycline in plasma, whole blood, dried blood spots (DBS), urine and hair after a single dose of doxycycline in men using oral doxycycline for post-exposure prophylaxis of sexually transmitted infections (syphilis or Chlamydia trachomatis) and having sex with men.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patient
* Men who have Sex with Men (MSM) on PrEP or HIV-infected patients
* Patients who have not taken doxycycline for at least 3 months
* No symptoms of bacterial STI infection (chlamydia, gonorrhea, Mycoplasma genitalium or syphilis).
* Documented history of bacterial STI infection within the past 12 months
* Having had a risky intercourse within 24 hours and at the latest within 72 hours and for which a prescription of doxycycline in a single dose of 200 mg has been made within the framework of his usual follow-up.
* Free, informed, written consent, signed by the person and the investigator at the latest on the day of inclusion and before any examination carried out within the framework of the study (article L1122-1-1 of the Public Health Code).
* Person affiliated or benefiting from a social security system (article L1121-11 of the Public Health Code)

Exclusion Criteria:

* Systemic treatment with retinoids (Acnetrait®, Procuta®, Curacné®, Contracné®, ....).
* Treatment with enzyme-inducing anticonvulsants (carbamazepine, phenobarbital, phenytoin, etc.).
* Known allergy to antibiotics of the tetracycline family.
* Known allergy to one of the components of doxycycline tablets.
* Documented esophageal injury
* Ongoing treatment with doxycycline at the time of inclusion.
* Person participating in another research study with an exclusion period still in progress at inclusion.
* Persons under guardianship, conservatorship, or deprived of liberty by judicial or administrative decision.
* Patients on State Medical Aid

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
Concentration of doxycycline in urine | At Day 90

SECONDARY OUTCOMES:
Concentration of doxycycline in plasma | Before the single intake of doxycycline
Concentration of doxycycline in plasma | 2 hours after doxycycline intake
Concentration of doxycycline in plasma | 24 hours after doxycycline intake
Concentration of doxycycline in plasma | 48 hours after doxycycline intake
Concentration of doxycycline in plasma | 7 days after doxycycline intake
Concentration of doxycycline in plasma | 14 days after doxycycline intake
Concentration of doxycycline in plasma | 30 days after doxycycline intake
Concentration of doxycycline in plasma | 60 days after doxycycline intake
Concentration of doxycycline in plasma | 90 days after doxycycline intake
Concentration of doxycycline in whole blood | Before the single intake of doxycycline
Concentration of doxycycline in whole blood | 2 hours after doxycycline intake
Concentration of doxycycline in whole blood | 24 hours after doxycycline intake
Concentration of doxycycline in whole blood | 48 hours after doxycycline intake
Concentration of doxycycline in whole blood | 7 days after doxycycline intake
Concentration of doxycycline in whole blood | 14 days after doxycycline intake
Concentration of doxycycline in whole blood | 30 days after doxycycline intake
Concentration of doxycycline in whole blood | 60 days after doxycycline intake
Concentration of doxycycline in whole blood | 90 days after doxycycline intake
Concentration of doxycycline in Dried Blood Spot (DBS) | Before the single intake of doxycycline
Concentration of doxycycline in Dried Blood Spot (DBS) | 2 hours after doxycycline intake
Concentration of doxycycline in Dried Blood Spot (DBS) | 24 hours after doxycycline intake
Concentration of doxycycline in Dried Blood Spot (DBS) | 48 hours after doxycycline intake
Concentration of doxycycline in Dried Blood Spot (DBS) | 7 days after doxycycline intake
Concentration of doxycycline in Dried Blood Spot (DBS) | 14 days after doxycycline intake
Concentration of doxycycline in Dried Blood Spot (DBS) | 30 days after doxycycline intake
Concentration of doxycycline in Dried Blood Spot (DBS) | 60 days after doxycycline intake
Concentration of doxycycline in Dried Blood Spot (DBS) | 90 days after doxycycline intake
Concentration of doxycycline in urine | Before the single intake of doxycycline
Concentration of doxycycline in urine | 2 hours after doxycycline intake
Concentration of doxycycline in urine | 24 hours after doxycycline intake
Concentration of doxycycline in urine | 48 hours after doxycycline intake
Concentration of doxycycline in urine | 7 days after doxycycline intake
Concentration of doxycycline in urine | 14 days after doxycycline intake
Concentration of doxycycline in urine | 30 days after doxycycline intake
Concentration of doxycycline in urine | 60 days after doxycycline intake
Concentration of doxycycline in urine | 90 days after doxycycline intake
Concentration of doxycycline in oropharyngeal secretions | Before the single intake of doxycycline
Concentration of doxycycline in oropharyngeal secretions | 2 hours after doxycycline intake
Concentration of doxycycline in oropharyngeal secretions | 24 hours after doxycycline intake
Concentration of doxycycline in oropharyngeal secretions | 48 hours after doxycycline intake
Concentration of doxycycline in oropharyngeal secretions | 7 days after doxycycline intake
Concentration of doxycycline in oropharyngeal secretions | 14 days after doxycycline intake
Concentration of doxycycline in oropharyngeal secretions | 30 days after doxycycline intake
Concentration of doxycycline in oropharyngeal secretions | 60 days after doxycycline intake
Concentration of doxycycline in oropharyngeal secretions | 90 days after doxycycline intake
Concentration of doxycycline in rectal secretions | Before the single intake of doxycycline
Concentration of doxycycline in rectal secretions | 2 hours after doxycycline intake
Concentration of doxycycline in rectal secretions | 24 hours after doxycycline intake
Concentration of doxycycline in rectal secretions | 48 hours after doxycycline intake
Concentration of doxycycline in rectal secretions | 7 days after doxycycline intake
Concentration of doxycycline in rectal secretions | 14 days after doxycycline intake
Concentration of doxycycline in rectal secretions | 30 days after doxycycline intake
Concentration of doxycycline in rectal secretions | 60 days after doxycycline intake
Concentration of doxycycline in rectal secretions | 90 days after doxycycline intake
Doxycycline concentration in hair | Before the single intake of doxycycline
Doxycycline concentration in hair | 1 month after doxycycline intake
Doxycycline concentration in hair | 3 months after doxycycline intake
Number of biological matrix(es) associated with a quantifiable doxycycline dosage | Up to 15 days
  Determine the biological matrix(es) associated with a quantifiable doxycycline dosage in more than 90% of the samples collected during the study.
Number of biological matrix(es) associated with a quantifiable doxycycline dosage | Up to 30 days
  Determine the biological matrix(es) associated with a quantifiable doxycycline dosage in more than 90% of the samples collected during the study.
Number of biological matrix(es) associated with a quantifiable doxycycline dosage | Up to 60 days
  Determine the biological matrix(es) associated with a quantifiable doxycycline dosage in more than 90% of the samples collected during the study.
Number of biological matrix(es) associated with a quantifiable doxycycline dosage | Up to 90 days
  Determine the biological matrix(es) associated with a quantifiable doxycycline dosage in more than 90% of the samples collected during the study.
Cmax (maximum concentration) in plasma | Until day 90
Cmax (maximum concentration) in whole blood | Until day 90
Cmax (maximum concentration) in Dried Blood Spot (DBS) | Until day 90
Cmax (maximum concentration) in urine | Until day 90
Cmax (maximum concentration) in hair | Until day 90
Cmax (maximum concentration) in rectal secretions | Until day 90
AUC (area under the curve) in plasma | Until day 90
AUC (area under the curve) in whole blood | Until day 90
AUC (area under the curve) in Dried Blood Spot (DBS) | Until day 90
AUC (area under the curve) in urine | Until day 90
AUC (area under the curve) in hair | Until day 90
AUC (area under the curve) in rectal secretions | Until day 90
Elimination clearance in plasma | Until day 90
Elimination clearance in whole blood | Until day 90
Elimination clearance in Dried Blood Spot (DBS) | Until day 90
Elimination clearance in urine | Until day 90
Elimination clearance in hair | Until day 90
Elimination clearance in rectal secretions | Until day 90
Half-life in plasma | Until day 90
Half-life in whole blood | Until day 90
Half-life in Dried Blood Spot (DBS) | Until day 90
Half-life in urine | Until day 90
Half-life in hair | Until day 90
Half-life in rectal secretions | Until day 90
Mean residence time in plasma | Until day 90
Mean residence time in whole blood | Until day 90
Mean residence time in Dried Blood Spot (DBS) | Until day 90
Mean residence time in urine | Until day 90
Mean residence time in hair | Until day 90
Mean residence time in rectal secretions | Until day 90
Volume of distribution in plasma | Until day 90
Volume of distribution in whole blood | Until day 90
Volume of distribution in Dried Blood Spot (DBS) | Until day 90
Volume of distribution in urine | Until day 90
Volume of distribution in hair | Until day 90
Volume of distribution in rectal secretions | Until day 90

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Lariboisière AP-HP, Paris
  - Hôpital Saint Louis AP-HP, Paris

IPD SHARING:
Plan to Share IPD: Undecided